CLINICAL TRIAL: NCT02748564
Title: Trial of Interleukin-2 in Combination With Pembrolizumab for Patients With Unresectable or Metastatic Melanoma
Brief Title: Aldesleukin and Pembrolizumab in Treating Patients With Stage III-IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study Complete
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Adam Berger, MD, Assistant Professor of Medicine Medical Oncology, Rutgers Cancer Institute of New Jersey
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 091602; NCI-2016-00466 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); Pro20160000394 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2016-04-19; First posted 2016-04-22 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Metastatic Melanoma; Stage III Mucosal Melanoma of the Head and Neck; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma; Stage IVA Mucosal Melanoma of the Head and Neck; Stage IVB Mucosal Melanoma of the Head and Neck; Stage IVC Mucosal Melanoma of the Head and Neck
MeSH Terms: conditions — Melanoma | interventions — aldesleukin; pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose escalation study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, aldesleukin) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1 every 3 weeks and aldesleukin IV every 8 hours for up to 14 doses at weeks 4, 7, 16, 19, 28, and 31 in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Aldesleukin; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Biological: Aldesleukin — Given IV
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This study will evaluate the safety and tolerability of IL-2 when given in combination with pembrolizumab to patients with advanced melanoma. Aldesleukin may stimulate white blood cells to melanoma cells. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Giving aldesleukin and pembrolizumab may kill more tumor cells.

There are two parts to this study:

* Phase Ib: To determine the safety and side effects of increasing doses of IL-2 in combination with pembrolizumab
* Phase II: Once the maximum tolerated dose of IL-2 is determined, additional patients will be treated to determine if it is effective against the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine an optimal tolerated dose (OTD) of aldesleukin (interleukin [IL]-2) that is effective and tolerable in combination with pembrolizumab.

II. To characterize the efficacy of the OTD of IL-2 in combination with pembrolizumab.

SECONDARY OBJECTIVES:

I. To characterize the safety of IL-2 in doses ranging up to the Food and Drug Administration (FDA)- approved dose when administered in combination with pembrolizumab.

II. To characterize clinical endpoints, including overall survival, progression-free survival, and complete response rate.

TERTIARY OBJECTIVES:

I. To characterize immune parameters in the blood and tumor microenvironment and cellular and molecular features of the tumor tissue that correlate with response to combination therapy for study as potential predictive biomarkers.

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1 every 3 weeks and aldesleukin IV every 8 hours for up to 14 doses at weeks 4, 7, 16, 19, 28, and 31 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of cutaneous melanoma, mucosal melanoma, or melanoma of unknown primary that is considered unresectable (stage III) or metastatic (stage IV)
* Be willing and able to provide written informed consent/assent for the trial
* Have measurable disease evident on radiographs (preferred) or clinical examination; for this protocol, measurable disease is defined as at least one evaluable tumor that is at least 10 mm in longest dimension
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Patients must have a brain magnetic resonance imaging (MRI) or computed tomography (CT) (with and without contrast) that is free of active metastases; metastases that have been treated with radiation or surgical resection, are stable for at least 4 weeks and do not require steroids are eligible
* Normal cardiac function; patients who have a history of heart disease, or who are over the age of 50 years must have a normal cardiac stress test within the prior 90 days
* Normal lung function; patients who have extensive pulmonary metastases or any chronic pulmonary disease history must have pulmonary function testing demonstrating forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) > 65% of predicted values
* Absolute neutrophil count (ANC) >= 1,500 /mcL
* Platelets >= 100,000 / mcL
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN OR =< 5 X ULN for subjects with liver metastases
* Albumin >= 2.5 mg/dL
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants
* Activated partial thromboplastin time (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication; subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy
* Subject meets institutional requirements for IL-2 therapy

Exclusion Criteria:

* Has primary ocular melanoma
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving systemic immunosuppressive steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of trial treatment; exception: physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency is not considered systemic immunosuppressive steroid therapy
* Has received previous high dose IL-2 therapy, any programmed death (PD)-1 blocking antibody (e.g. pembrolizumab, nivolumab), or any programmed death ligand (PD-L)1 blocking antibody in the metastatic setting; prior therapy with any PD-1 blocking antibody is allowed if given in the adjuvant setting and the last dose was > 6 months prior to study entry; prior therapy with ipilimumab is allowed (in the adjuvant or metastatic setting); other prior therapy (in the adjuvant or the metastatic setting) is allowed, including targeted therapy, chemotherapy, or experimental therapy
* Has a history of significant congestive heart failure or significant pulmonary disease
* Has a known history of active TB (bacillus tuberculosis)
* Hypersensitivity to pembrolizumab or any of its excipients
* Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: subjects with =< grade 2 neuropathy and/or alopecia are exceptions to this criterion and may qualify for the study
  * Note: if subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis; subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Has known history of, or any evidence of active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies)
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days of planned start of study therapy

  * Note: seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-10-18 (Actual); Study Completion 2023-06-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Berger, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (5):
- United States (5):
  - Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Indiana University, Bloomington, Indiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Silk AW, Curti B, Bryan J, Saunders T, Shih W, Kane MP, Hannon P, Fountain C, Felcher J, Zloza A, Kaufman HL, Mehnert JM, McDermott DF. A phase Ib study of interleukin-2 plus pembrolizumab for patients with advanced melanoma. Front Oncol. 2023 Feb 9;13:1108341. doi: 10.3389/fonc.2023.1108341. eCollection 2023. PMID 36845705

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All collected data for pre-specified Primary and Secondary Outcome Measures, and accurate Participant Flow, Baseline, and Adverse Events data is expected to be reported. Funding was lost so the second half of the study could not be completed.
Groups:
- Level 1 Treatment Pembrolizumab 200mg IV IL-2 6,000: Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 6,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
- Level 2 Pembrolizumab 200mg IV IL-2 60,000: Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 60,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
- Level 3 Pembrolizumab 200mg IV IL-2 600,000: Experimental 600,000 IU/kg of IL -2
  Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 600,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
Period: Overall Study
Arm/Group | Level 1 Treatment Pembrolizumab 200mg IV IL-2 6,000 | Level 2 Pembrolizumab 200mg IV IL-2 60,000 | Level 3 Pembrolizumab 200mg IV IL-2 600,000
Started | 3 | 3 | 4
Completed | 3 | 3 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Level 1 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 6,000: Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 6,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
- Level 2 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 60,000z: Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 60,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
- Level 3 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 600,000: Additionally, participants receive IL-2 6,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
- Total: Total of all reporting groups
Arm/Group | Level 1 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 6,000 | Level 2 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 60,000z | Level 3 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 600,000 | Total
Number analyzed (Participants) | 3 | 3 | 4 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 3 | 8
  >=65 years | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 4
  Male | 1 | 2 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 3 | 3 | 4 | 10
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate as Assessed by Response (BORR) Evaluation Criteria in Solid Tumors Version 1.1, With the Modification That Progressive Disease Must be Confirmed on a Subsequent Scan
Description: Estimated using OTD of IL-2 and pembrolizumab assessed by Response Evaluation Criteria in Solid Tumors version 1.1,for target lesions and assessed by CT or MRI imaging: Complete response (CR) - disappearance of all target lesions; Partial response (PR) - >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) - At least a 20% increase in the sum of the longest diameter of target lesions; or Stable Disease (SD) - neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  By testing increasing doses up to 600,000 IU. Receive IL-2 6,000 International Units per kilogram (IU/kg);in cycles 2, 3, 6,7,10 and 11, with follow up thirty days after the last dose of study drug
Time Frame: Four to six weeks later up to one year
Measure: Count of Participants; unit: Participants
Groups:
- Level 1 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 6,000 Aldesleukin): Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 6,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
- Level 2 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 60,000: Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 60,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
Arm/Group | Level 1 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 6,000 Aldesleukin) | Level 2 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 60,000 | Level 3 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 600,000
Number analyzed (Participants) | 3 | 3 | 4
Participants | 0 | 0 | 0

2. Secondary Outcome: Complete Response Rate
Description: Participants are treated with pembrolizumab and the MTD of IL-2. Will be measured using the RECIST v 1.1. For all participants who experience a complete response, the date noted for disease response is the time of the scan when it was originally determined, and not the later date of the confirmatory scan.
Time Frame: Four to six weeks later, up to three years
Population: The Number of Participants Analyzed for each Row should be specified in the Number Analyzed row, since it differs from the Overall Number of Participants Analyzed specified.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Aldesleukin)
Number analyzed (Participants) | 10
Participants
  Level 1: number analyzed (Participants) | 3
  Level 1 | 0
  Level 2: number analyzed (Participants) | 3
  Level 2 | 0
  Level 3: number analyzed (Participants) | 4
  Level 3 | 1

3. Secondary Outcome: Number of Adverse Effects (AE) as Evaluated by National Cancer Institute Common Terminology Criteria for AE's, Version 4.0
Description: Each participant will be assessed for potential or new worsening AE's. AE's will be graded and recorded through the study and during follow-up period according to National Cancer Institute Common Terminology Criteria for AE's, version 4.0. Grade 1-5 with grade 5 being the most severe.
Time Frame: Thirty days after last dose of treatment, up to three years
Population: The Number of Participants Analyzed for each Row should be specified, since it differs from the Overall Number of Participants Analyzed specified.
Measure: Number; unit: Grade 3 or higher AE's
Arm/Group | Treatment (Pembrolizumab, Aldesleukin)
Number analyzed (Participants) | 10
Grade 3 or higher AE's
  Level 1: number analyzed (Participants) | 3
  Level 1 | 0
  Level 2: number analyzed (Participants) | 3
  Level 2 | 2
  Level 3: number analyzed (Participants) | 4
  Level 3 | 3

4. Secondary Outcome: Overall Survival Estimated Using Kaplan-Meier Curves
Description: Assess for survival status until death. Time to death measured in months.
Time Frame: Baseline to end of follow-up, up to 3 years
Population: as for outcome 3
Measure: Mean (Full Range); unit: months
Arm/Group | Treatment (Pembrolizumab, Aldesleukin)
Number analyzed (Participants) | 10
months
  Level 1: number analyzed (Participants) | 3
  Level 1 | 20.4 [4 to 56]
  Level 2: number analyzed (Participants) | 3
  Level 2 | 20.4 [4 to 56]
  Level 3: number analyzed (Participants) | 4
  Level 3 | 20.4 [4 to 56]

5. Secondary Outcome: Progressive Free Survival Retaining Progression-free Survival Status up to 36 Months
Description: As measured by Response Evaluation Criteria in Solid Tumors (RECIST v1.1) for targeted lesions; Partial response (PR) - >= 30% increase in the sum of the longest diameter of target lesions; or stable (SD) - neither sufficient shrinkage to quality for PR nor Sufficient increase to quality PD. Descriptive statistical will be used. Continuous variables will be presented by summary statistics (such as mean, median, standard error and 90% CI) and the categorical variables by frequency distributions (i.e., frequency counts, percentages and 90% CI).
Time Frame: Up to three years
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab, Aldesleukin)
Number analyzed (Participants) | 10
Participants
  Level 1: number analyzed (Participants) | 3
  Level 1 | 0
  Level 2: number analyzed (Participants) | 3
  Level 2 | 0
  Level 3: number analyzed (Participants) | 4
  Level 3 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after last dose of treatment and up to three years.
Groups:
- Level 1 Treatment Pembrolizumab 200mg IV Q3 wk, IL-2 6,000: Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 6,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
- Level 3 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 600,000: Cohort 1: Participants were administered 200mg of Pembrolizumab by an infusion into a vein or central line every three weeks. The infusion time is 30 minutes.
  Additionally, participants receive IL-2 600,000 International Units per kilogram (IU/kg); in cycles 2, 3, 6,7,10 and 11, with follow up 30 days after the last dose of study drug.
  Participants will receive Pembrolizumab first followed by IL-2 every 8 hours up to a total of 14 doses.
Arm/Group | Level 1 Treatment Pembrolizumab 200mg IV Q3 wk, IL-2 6,000 | Level 2 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 60,000 | Level 3 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 600,000
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 4/4
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 4/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 Treatment Pembrolizumab 200mg IV Q3 wk, IL-2 6,000 (N=3) | Level 2 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 60,000 (N=3) | Level 3 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 600,000 (N=4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Level 1 Treatment Pembrolizumab 200mg IV Q3 wk, IL-2 6,000 (N=3) | Level 2 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 60,000 (N=3) | Level 3 Treatment Pembrolizumab 200mg IV Q3 wk IL-2 600,000 (N=4)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) | 1 (2) | 1 (2)
General Disorders (General disorders) | 3 (8) | 3 (4) | 3 (6)
Infections (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Gastro disorder (Gastrointestinal disorders) | 3 (4) | 2 (8) | 2 (7)
Investigations (Investigations) | 2 (3) | 2 (16) | 3 (21)
Metabolism (Metabolism and nutrition disorders) | 1 (2) | 2 (11) | 2 (7)
Psychiatic (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (10)
Renal (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3) | 2 (6)
Vascular (Vascular disorders) | 1 (2) | 1 (1) | 1 (3)
Muscular Skeleton (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 1 (1)
Respirtory (Respiratory, thoracic and mediastinal disorders) | 1 (7) | 1 (1) | 3 (12)
Reproductive (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Immune (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Blood (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Protocol SAP #2 (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02748564/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: Protocol SAP #3 (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02748564/Prot_SAP_002.pdf
  • Statistical Analysis Plan: Protocol SAP #1 (2021-09-21): https://cdn.clinicaltrials.gov/large-docs/64/NCT02748564/SAP_003.pdf